CLINICAL TRIAL: NCT03666689
Title: Outflow Reconstruction in Right Lobe Living Donor Liver Transplantation: Middle Hepatic Vein Reconstruction Versus Separate Tributaries to Inferior Vena Cava Anastomosis
Brief Title: Outflow Reconstruction in Right Lobe Living Donor Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abdalla, assisstant lecturer, Assiut University
Other Study IDs: MHV reconstruction in LDLT
Record Dates: First submitted 2018-09-09; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Liver Transplant
MeSH Terms: interventions — Wound Closure Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MHV reconstruction: Both ends of middle hepatic vein tributaries V8 and/or V5 of modified right lobe graft will be anastomosed to side of a single synthetic graft which will be anastomosed to recipient's middle/left hepatic vein orifice.
  Interventions: Procedure: surgical technique
- Separate tributaries reconstruction: End of V8 middle hepatic vein tributary of modified right lobe graft; if present, will be anastomosed to end of a synthetic graft which will be anastomosed to recipient's middle/left hepatic vein orifice, and end of V5; if present; will be anastomosed to end of a synthetic graft which will be anastomosed to recipient's Inferior Vena Cava directly.
  Interventions: Procedure: surgical technique

INTERVENTIONS:
Procedure: surgical technique — surgical reconstruction

SUMMARY:
Modified Right Lobe Graft(MRLG) is one of the most common used graft in liver transplantation .Anterior sector of allograft in MRLG usually congested to decrease this congestion tributaries of middle hepatic vein should be drained to inferior vena cava .

There are too many techniques available for this drainage using either cryopreserved or synthetic graft for vascular anastomosis .In this study we will compare between two different technique using ringed synthetic polytetrafluoroethylene (PTFE) graft to assess outflow adequacy in both technique.

DETAILED DESCRIPTION:
Comparative, prospective, observational, two-groups study. group 1 : Middle Hepatic Vein(MHV) will reconstructed by fashioning a PTFE graft of suitable size positioned parallel to the cut surface of the Modified Right Lobe Graft.This position theoretically make the PTFE graft in a position similar to MHV.Any vein >4mm will be connected end to side fashion to the PTFE graft.The distal end of the PTFE graft will be closed by hemolock just distal to segment 5 vein .The proximal end of PTFE graft will be anastomosed to the recipient MHV orifice or MHV/lift orifice group 2: The end of segment 5 vein will be anastomosed to the end of suitable size PTFE graft which will be anastomosed to Inferior Vena Cava (IVC) directly and The end of segment 8 vein will be anastomosed to the end of suitable size PTFE graft which will be anastomosed to MHV or MHV/Lift orifice directly.the study will not be randomized .All operation will be done by tha same team .Choice of technique at surgeon discretion .Outflow adequecy will be assessed by Doppler Ultrasound intraoperatively and daily for 5 day once per week for 4 week and ,2,3,6,month.Progressive diminished flow or absent flow both will be considered as graft not patent .Markers of venous congestion will be considered as secondary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing Living Donor Liver Transplantation(LDLT) accepted according to hospital protocol
* Written informed consent obtained
* patient undergoing venous reconstruction either segment 5 or segment 8 vein or both

Exclusion Criteria:

* Acute fulminant liver failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will included in the study all patients accepted for Living Donor Liver Transplantation (LDLT) according to hospital protocol
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Outflow adequacy of liver graft within the first 6 month post transplant | 6 month
  Outflow adequacy of the graft will be assessed intraoperatively by the presence of the congestion and the color of the graft and Doppler ultrasound will be done after vascular reconstruction and before closure of anterior abdominal wall. Outflow adequacy will be assessed postoperatively by Doppler ultrasound once per day for the first 5 days, then once per week for 4 weeks then 2,3,and 6 months. Computed tomography (CT) scan will be done in the 6 postoperative month

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lo CM, Fan ST, Liu CL, Wei WI, Lo RJ, Lai CL, Chan JK, Ng IO, Fung A, Wong J. Adult-to-adult living donor liver transplantation using extended right lobe grafts. Ann Surg. 1997 Sep;226(3):261-9; discussion 269-70. doi: 10.1097/00000658-199709000-00005. PMID 9339932
- [Background] Fan ST, Lo CM, Liu CL, Wang WX, Wong J. Safety and necessity of including the middle hepatic vein in the right lobe graft in adult-to-adult live donor liver transplantation. Ann Surg. 2003 Jul;238(1):137-48. doi: 10.1097/01.sla.0000077921.38307.16. PMID 12832976
- [Background] Yi NJ, Suh KS, Lee HW, Cho EH, Shin WY, Cho JY, Lee KU. An artificial vascular graft is a useful interpositional material for drainage of the right anterior section in living donor liver transplantation. Liver Transpl. 2007 Aug;13(8):1159-67. doi: 10.1002/lt.21213. PMID 17663413
- [Background] Hwang S, Jung DH, Ha TY, Ahn CS, Moon DB, Kim KH, Song GW, Park GC, Jung SW, Yoon SY, Namgoong JM, Park CS, Park YH, Park HW, Lee HJ, Lee SG. Usability of ringed polytetrafluoroethylene grafts for middle hepatic vein reconstruction during living donor liver transplantation. Liver Transpl. 2012 Aug;18(8):955-65. doi: 10.1002/lt.23456. PMID 22511404